CLINICAL TRIAL: NCT01308281
Title: Impact of IntraVascular UltraSound Guidance on Outcomes of Xience Prime Stents in Long Lesions (IVUS-XPL Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2010-0025
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI with IVUS guidance (Experimental): PCI(percutaneous coronary intervention) with IVUS(IntraVascular UltraSound) group
  Interventions: Procedure: PCI with IVUS guidance
- PCI without IVUS guidance (Active Comparator): PCI(percutaneous coronary intervention) group
  Interventions: Procedure: PCI without IVUS guidance

INTERVENTIONS:
Procedure: PCI with IVUS guidance — Patients will be randomized in a two-by-two factorial manner according to the use of IVUS guidance (IVUS guidance vs. no IVUS guidance) for the PCI and the duration of dual anti-platelet therapy (100 mg/day aspirin and 75mg/day clopidogrel for 6 months vs. 12 months) after PCI. Each randomization of the enrolled subjects will be done 1:1.
  Other Names: PCI with IVUS guidance group
  Arms: PCI with IVUS guidance
Procedure: PCI without IVUS guidance — Patients will be randomized in a two-by-two factorial manner according to the use of IVUS guidance (IVUS guidance vs. no IVUS guidance) for the PCI and the duration of dual anti-platelet therapy (100 mg/day aspirin and 75mg/day clopidogrel for 6 months vs. 12 months) after PCI. Each randomization of the enrolled subjects will be done 1:1.
  Arms: PCI without IVUS guidance

SUMMARY:
This study is designed as a prospective, randomized, multi-center trial to demonstrate an inequality between IVUS-guided versus angiography-guided implantation of everolimus-eluting stents(EES) at long lesions(> 28 mm) in clinical outcomes at 12 months as a primary objective and safety of 6- month dual antiplatelet therapy following EES implantation in comparison with a 12-month dual antiplatelet therapy.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate the impact of IVUS guidance on the clinical outcomes after implantation of DES at long lesions > 28 mm.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years old or older
* Patients with typical chest pain or evidences of myocardial ischemia (e.g., stable, unstable angina, silent ischemia and positive functional study or reversible changes in the electrocardiogram (ECG) consistent with ischemia
* Non-emergent conditions
* Patients with signed informed consent
* Stent length ≥28 mm by angiography estimation
* Significant coronary artery stenosis (> 50% by visual estimate) considered for coronary revascularization with stent implantation
* Reference vessel diameter of 2.5 to 4.0 mm by operator assessment

Exclusion Criteria:

* Acute ST elevation myocardial infarction within 48 hours
* Contraindication to anti-platelet agents & bleeding history within prior 3 months
* Known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Zotarolimus or other -limus group
* Prior history of the following presentations

  * Cerebral vascular accident (not including transient ischemic attack)
  * Peripheral artery occlusive diseases
  * Thromboembolic disease
  * Stent thrombosis
* Age > 80 years old
* Severe hepatic dysfunction (3 times normal reference values)
* Significant renal dysfunction (Serum creatinine > 2.0 mg/dl)
* Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* Cardiogenic shock
* LVEF < 40%
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year
* Left main disease requiring PCI
* Bifurcation lesion with 2-stent technique
* Chronic total occlusion
* Presence of previously implanted DES within 6-month
* In-stent restenosis lesion

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1079 (Actual)
Dates: Start 2010-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event, a composite of cardiac death, target lesion related MI, target lesion revascularization following randomly assigned PCI procedures with versus without IVUS guidance | 12 months after the index procedure
  Major adverse cardiac event, a composite of cardiac death, target lesion related MI, target lesion revascularization following randomly assigned PCI procedures with versus without IVUS guidance

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jin IT, Kim Y, Heo SJ, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Kim JS, Cho DK, Ko YG, Choi D, Hong MK, Kim BK. Comparison of Short-term and Standard Duration Dual Antiplatelet Therapy in Elderly Patients: A Pooled Analysis of Five Korean Randomized Clinical Trials. Korean Circ J. 2025 Dec;55(12):1125-1137. doi: 10.4070/kcj.2025.0093. Epub 2025 Jul 14. PMID 41044734
- [Derived] Lee SY, Zhang JJ, Mintz GS, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Kan J, Pan T, Gao X, Ge Z, Chen SL, Hong MK. Procedural Characteristics of Intravascular Ultrasound-Guided Percutaneous Coronary Intervention and Their Clinical Implications. J Am Heart Assoc. 2022 Jul 19;11(14):e025258. doi: 10.1161/JAHA.122.025258. Epub 2022 Jul 15. PMID 35861828
- [Derived] Jang JY, Jung HW, Lee BK, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Kwon HM, Jang Y. Impact of PRECISE-DAPT and DAPT Scores on Dual Antiplatelet Therapy Duration After 2nd Generation Drug-Eluting Stent Implantation. Cardiovasc Drugs Ther. 2021 Apr;35(2):343-352. doi: 10.1007/s10557-020-07008-7. PMID 32588238
- [Derived] Jang JY, Shin DH, Kim JS, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Park KW, Gwon HC, Kim HS, Jang Y. Optimal duration of DAPT after second-generation drug-eluting stent in acute coronary syndrome. PLoS One. 2018 Nov 26;13(11):e0207386. doi: 10.1371/journal.pone.0207386. eCollection 2018. PMID 30475845
- [Derived] Hong SJ, Shin DH, Kim JS, Kim BK, Ko YG, Choi D, Her AY, Kim YH, Jang Y, Hong MK; IVUS-XPL Investigators. 6-Month Versus 12-Month Dual-Antiplatelet Therapy Following Long Everolimus-Eluting Stent Implantation: The IVUS-XPL Randomized Clinical Trial. JACC Cardiovasc Interv. 2016 Jul 25;9(14):1438-46. doi: 10.1016/j.jcin.2016.04.036. Epub 2016 May 17. PMID 27212028
- [Derived] Hong SJ, Kim BK, Shin DH, Nam CM, Kim JS, Ko YG, Choi D, Kang TS, Kang WC, Her AY, Kim YH, Hur SH, Hong BK, Kwon H, Jang Y, Hong MK; IVUS-XPL Investigators. Effect of Intravascular Ultrasound-Guided vs Angiography-Guided Everolimus-Eluting Stent Implantation: The IVUS-XPL Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2155-63. doi: 10.1001/jama.2015.15454. PMID 26556051